CLINICAL TRIAL: NCT02793115
Title: Physician Disclosures in the Real World of Conflicting Interests
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Susannah Rose, Associate Staff, The Cleveland Clinic
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 14-1438
Record Dates: First submitted 2016-06-03; First posted 2016-06-08 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Conflicts of Interest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm 1 (Experimental): Disclosure Letter-RISKS
  Interventions: Behavioral: Disclosure Letter-RISKS
- Arm 2 (Experimental): Disclosure Letter-BENEFITS
  Interventions: Behavioral: Disclosure Letter-BENEFITS
- Arm 3 (Experimental): Disclosure Letter-RISKS AND BENEFITS
  Interventions: Behavioral: Disclosure Letter-RISKS AND BENEFITS
- Arm 4 (Experimental): Disclosure Letter-NO RISKS OR BENEFITS
  Interventions: Behavioral: Disclosure Letter-NO RISKS OR BENEFITS
- Arm 5 (Placebo Comparator): Letter-APPOINTMENT REMINDER
  Interventions: Behavioral: Letter-APPOINTMENT REMINDER

INTERVENTIONS:
Behavioral: Disclosure Letter-RISKS — This disclosure letter will provide information on the physicians' financial relationships with industry, and will also provide a standardized statement regarding the potential RISKS of physicians' conflicts of interest with for-profit industry. This letter also includes a standard statement reminding the patient about the appointment and the location of the appointment.
  Arms: Arm 1
Behavioral: Disclosure Letter-BENEFITS — This disclosure letter will provide information on the physicians' financial relationships with industry, and will also provide a standardized statement regarding the potential BENEFITS of physicians' conflicts of interest with for-profit industry. This letter also includes a standard statement reminding the patient about the appointment and the location of the appointment.
  Arms: Arm 2
Behavioral: Disclosure Letter-RISKS AND BENEFITS — This disclosure letter will provide information on the physicians' financial relationships with industry, and will also provide a standardized statement regarding the potential RISKS AND BENEFITS of physicians' conflicts of interest with for-profit industry. This letter also includes a standard statement reminding the patient about the appointment and the location of the appointment.
  Arms: Arm 3
Behavioral: Disclosure Letter-NO RISKS OR BENEFITS — This letter includes a standard statement reminding the patient about the appointment and the location of the appointment.and DOES NOT provide any information on the physicians' financial relationships with industry nor information regarding the potential risks and benefits of physicians' conflicts of interest with for-profit industry.
  Arms: Arm 4
Behavioral: Letter-APPOINTMENT REMINDER — This letter only includes a standard statement reminding the patient about the appointment and the location of the appointment.
  Arms: Arm 5

SUMMARY:
This study seeks to ascertain the best way to inform patients about their physicians' conflicts of interest (COI) with industry. Currently, there is no institutional or national standard for such physician-to-patient disclosures. The primary aim of this study is to test different written disclosures and assess their impact on patients' knowledge of their physicians' COIs and on patients' trust in their physician and their healthcare institution. The secondary aim is to investigate whether physician disclosures of significant financial industry relationships are desired by patients and whether disclosures impact patients' knowledge, perceptions, and behaviors. The tertiary aim is to investigate physicians' current practices of disclosure and perceptions about the risks, benefits, and feasibility of using patient disclosures to manage financial relationships, and to determine whether any physician fears are borne out in practice once disclosures are implemented.

DETAILED DESCRIPTION:
This study uses a mixed-methods design. A randomized intervention (RCT) will be a mailed letter sent to approximately 1310 patients, disclosing their physicians' financial relationships with industry before patients meet with their physicians. There are 4 experimental conditions, systematically varying the wording of the COI disclosures, and one control condition. These patients will be briefly surveyed after they see their physicians, using standardized measures of trust and other questions. The goal is to achieve a 65% response rate (final n=850).

The sample size was determined based on a 0.3 unit change in Mayer Trust Scale adapted to refer to "physician" rather than "management" between the subgroups using the POWER procedure in SAS software version 9.3. In its original presentation, the Mayer Trust Scale lists a standard deviation for the 4-item trust score as 0.66 - 0.68. A sample size of 850 patients (170 in each of the 5 groups) would provide 82% power to detect a 0.3 unit difference in Mayer Trust Scale after Bonferroni correction for the 10 possible comparisons, assuming a standard deviation of 0.7 and that the significance level of 0.005 (0.05 / 10 comparisons) would be used in these analyses. In addition, this sample size would allow for multivariable regression models sufficient parameters to be fit following the suggested ratio of 10 patients for each predictor in the model.

Additionally, to supplement patient-derived RCT survey results, approximately 25 Cleveland Clinic physicians with industry relationships over $20,000 will be interviewed to gather their perspectives on COI disclosure. These interviews will occur before and after the RCT, and will collect qualitative and quantitative data. Qualitative data will be analyzed using content analysis, an iterative process of data immersion and data coding, whereby narrative data is categorized into discrete codes based on thematic content and then used to compute descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

* Cleveland Clinic patients who have an appointment scheduled with a physician who receives at least $20,000 per year from a drug and device company.
* Patient's primary language is English.

Exclusion Criteria:

* Patients under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 895 (Actual)
Dates: Start 2014-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Patient Trust in Physician | Within approximately 1 month of intervention
  Self-reported trust in physicians, as assessed by standardized survey instrument.
Patient Trust in Hospital | Within approximately 1 month of intervention
  Self-reported trust in hospital, as assessed by standardized survey
Accuracy of Patient Knowledge of their Physicians' Industry Relationships | Within approximately 1 month of intervention
  Self-reported, assessed by survey questions.

REFERENCES:
- [Background] Gordon HS, Street RL Jr, Sharf BF, Kelly PA, Souchek J. Racial differences in trust and lung cancer patients' perceptions of physician communication. J Clin Oncol. 2006 Feb 20;24(6):904-9. doi: 10.1200/JCO.2005.03.1955. PMID 16484700
- [Background] Mayer RC, Davis JH, Schoorman FD. An integrative model of organizational trust. The Academy of Management Review 20(3): 709-734, 1995.